CLINICAL TRIAL: NCT00992888
Title: Inflammation, Immune Activation and Portal Hypertension in Alcoholic Hepatitis. A Pato-etiological Study With Focus on the Endotoxin Pathway.
Brief Title: Inflammation, Immune Activation and Portal Hypertension in Alcoholic Hepatitis
Acronym: Heliac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Thomas Damgaard Sandahl, Dr, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Heliac-01
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; Alcohol; Endotoxin; LPS; Liver dialysis; Innate immunity; Toll Like receptors
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- albumin liver dialysis (Experimental)
  Interventions: Device: Prometheus Liver Dialysis system (Fresenius Medical Care)
- Standard medial care without dialysis (No Intervention)

INTERVENTIONS:
Device: Prometheus Liver Dialysis system (Fresenius Medical Care) — 6 hour dialysis for 3 consecutive days
  Other Names: The prometheus albumin dialysis by Fresenius Medical Care
  Arms: albumin liver dialysis

SUMMARY:
The purpose of this study is to investigate the role of endotoxins and the endotoxin mediated immune activation pathway in patients with alcoholic hepatitis. Also, to determine the effect of Liver assist (liver dialyses) intervention on these parameters in patients with severe alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

Patients with alcoholic hepatitis based on the following criteria

* Alcohol intake for 6 consecutive months above 40g /day, at admission or 3 months earlier.
* Serum bilirubin level above 80 mmol/l
* exclusion of other types of liver disease.
* Liver biopsy when diagnosis is unclear.

Exclusion Criteria:

* Heart failure
* Pregnancy
* non fluent danish speakers

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Serum endotoxin levels | one year

SECONDARY OUTCOMES:
Endotoxin activation pathway proteins | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Vilstrup, Prof, Study Director — Department of Medicine V, Aarhus University Hospital
Locations (1):
- Department of Medicine V, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Stoy S, Dige A, Sandahl TD, Laursen TL, Buus C, Hokland M, Vilstrup H. Cytotoxic T lymphocytes and natural killer cells display impaired cytotoxic functions and reduced activation in patients with alcoholic hepatitis. Am J Physiol Gastrointest Liver Physiol. 2015 Feb 15;308(4):G269-76. doi: 10.1152/ajpgi.00200.2014. Epub 2014 Dec 11. PMID 25501547